CLINICAL TRIAL: NCT05018000
Title: CAFÉ: Clinic Based Intervention to Address Financial Hardship for People With Cancer
Brief Title: Cancer Financial Experience
Acronym: CAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1R01CA237322 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: financial hardship; cancer; health outcomes
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Enhanced usual care (Active Comparator): Participants in this arm will receive their usual care plus a Financial Resource Sheet. The financial resource sheet lists and describes existing organization and community resources available to KP members.
  Interventions: Behavioral: Enhanced usual care
- Arm 2: Brief financial navigation intervention (Experimental): Participants in this arm will receive their usual care, and the Financial Resource Sheet described in Arm 1, plus one (1) cycle of financial navigation (total cycles: 1; total length: 6 months). In each intervention cycle participants will get at least one (1) phone call with a CAFÉ Financial Navigator, the navigator will talk with participants to identify financial questions or concerns. The navigator will create a personalized plan for each participant. Participants can request extra support from the navigator for up to 6 months.
  Interventions: Behavioral: Financial navigation
- Arm 3: Extended financial navigation intervention (Experimental): Participants in this arm will receive their usual care, a Financial Resource Sheet and the brief intervention described in Arm 2 (i.e., one (1) cycle of financial navigation). Plus, they will receive two (2) additional cycles of financial navigation (total cycles: 3; total length: 6 months).
  Interventions: Behavioral: Financial navigation

INTERVENTIONS:
Behavioral: Financial navigation — The CAFÉ intervention is a financial navigation intervention. During the Intervention, a CAFÉ financial navigator will provide information support and resources to people with cancer after diagnosis. CAFÉ intervention components include: (1) proactive assessment of patient financial questions and concerns (e.g., acute financial need or inability to pay for household expenses; deciding between care options depending on cost; uncertainty around planning for out of pocket costs and/or when patients will need to pay), (2) proactive, personalized support and referrals.
  Arms: Arm 2: Brief financial navigation intervention; Arm 3: Extended financial navigation intervention
Behavioral: Enhanced usual care — The financial resource sheet lists and describes existing internal and community resources available to KP members
  Arms: Arm 1: Enhanced usual care

SUMMARY:
This study is a randomized clinical trial designed to test a novel financial navigation intervention. The study assesses the impact of the financial navigation intervention on financial hardship and health-related quality of life, cancer-related material and psychological financial hardship, patient-centered communication, and time to initiation of treatment.

DETAILED DESCRIPTION:
Rationale:

Up to half of people with cancer experience financial hardship. Cancer-related financial hardship is associated with several adverse intermediate and health outcomes, including poor quality of life, treatment non-adherence, and lower survival.

Observational evidence suggests that communication about financial concerns and out-of-pocket (OOP) costs early in the treatment trajectory and in partnership with the care team could help to prevent or lessen financial hardship. This type of communication could be delivered through patient navigation programs and is consistent with both patient and care team preferences.

However, to date there is no evidence from randomized trials showing the impact of financial navigation during the active treatment on financial hardship. Further, no intervention-based studies have provided evidence on the most effective ways to mitigate cancer-related financial hardship.

Background:

As costs of cancer care in U.S. have risen over time, so has the burden of out-of-pocket (OOP) costs and indirect costs such as travel, employment changes, and caregiver costs. These cumulative costs pose increased financial risk for people diagnosed with cancer. Despite a patient's health insurance status, financial hardship from cancer care is prevalent: 47%-49% of cancer survivors report financial hardship and 12%-62% of cancer survivors report debt due to treatment costs. Financial hardship is associated with decreased treatment initiation and adherence, poor symptoms and quality of life, and increased mortality risk, so preventing or mitigating its effects is a clinical imperative.

Integration of cost of cancer care information into conversations between patients and clinicians can optimize medical decision-making and reduce the risk of financial hardship, and is consistent with high-quality cancer care and patient preferences. Patient understanding of OOP costs can assist with planning and budgeting, and can facilitate early connection with financial support services that may help to mitigate the financial burden of cancer care. Yet, less than one in five patients report having cost discussions. Consequently, many patients are uninformed about the costs of their cancer care and face unexpected OOP costs, with important consequences for material (e.g., debt), psychological (e.g., cost-related distress), and behavioral (e.g. treatment adherence) financial hardship.

There is an urgent need for evidence-based interventions on how to prevent or mitigate financial hardship for people with cancer. While the extent of financial hardship as a toxicity of cancer care is increasingly well-documented, there is limited evidence to date as to what types of interventions can mitigate or prevent financial hardship due to cancer care. Policy, societal, and organizational-level interventions, such as those focused on bending the curve of rising health care cost or improving price transparency to ordering providers are all needed, but these may take a long time or show limited effect. In the meantime, patients continue to need assistance navigating, managing and anticipating OOP costs, and patient- and team level-interventions such as the CAFÉ study may hold promise for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. KPNW and KPWA members with a new cancer diagnosis (within the past 120 days from identification date)
2. 18+ years of age (based on age at time of identification date)
3. Recent visit to CAFÉ clinic/department
4. Current, living member as of identification date
5. Continuous enrollment at least 6 months prior to identification date
6. English speaker for KPWA; English or Spanish speaker for KPNW

Exclusion Criteria:

1. On do-not contact list at KP
2. Cancer diagnosis is for non-melanoma skin cancer
3. Cancer diagnosis is for a benign or in situ tumor
4. Hospice referral in past year
5. Self or household member has already enrolled or completed participation in CAFÉ pilot study or main trial.
6. Unable to complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Financial distress | baseline and 12 months
  InCharge Financial Distress/Financial Well-Being Scale. This is a validated, 8-item scale that assesses current ability to meet financial obligations, stress or worry about finances, and satisfaction with present financial situation. It is scored to a 10-point scale, where 1 is "Overwhelming financial distress/lowest financial well-being," and 10 is "No financial distress/highest financial well-being." It has been validated in multiple populations and national norms are provided.
Health-related quality of life (cancer specific) | baseline and 12 months
  The FACT-G7 is a 7-item version of the Functional Assessment of Cancer Therapy-General (FACT-G), a patient-reported outcome measure used to assess health-related quality of life in patients undergoing cancer therapy. The survey assesses the impacts of cancer therapy in four domains: physical, social/family, emotional, and functional. Higher scores represent higher quality of life.

SECONDARY OUTCOMES:
Financial hardship due to cancer care costs | baseline and 12 months
  Items from the Medical Expenditure Panel Survey (Yabroff 2016):
  Material financial hardship items:
  Have you or has anyone in your family had to borrow money or go into debt because of your cancer, its treatment or the lasting effects of that treatment? (Yes\No)
  Did you or your family ever file for bankruptcy because of your cancer, its treatment, or the lasting effects of that treatment? (Yes\No)
  Have you or your family had to make any other kinds of financial sacrifices because of your cancer, its treatment, or the lasting effects of that treatment? (Yes\No)
  Please think about medical care visits for cancer, its treatment, or the lasting effects of that treatment. Have you ever been unable to cover your share of those visits? (Yes\No)
  Psychological financial hardship item:
  Have you ever worried about having to pay large medical bills related to your cancer? (Yes\No)

OTHER OUTCOMES:
Initiation of cancer treatment | between baseline and 12 months
  Proportion of patients initiating treatment, including radiation, surgery, and systemic therapy.
Time to initiation of cancer treatment | between baseline and 12 months
  Defined as the number of days between: 1) date of diagnosis/recurrence and start of first-line treatment. Censoring events will include disenrollment, death, and end of the study, whichever comes first.
Use of medical financial assistance (MFA) | between baseline and 12 months
  Proportion of participants who enrolled in the Kaiser Permanente MFA program within 12 months following baseline
Delinquent account | between baseline and 12 months
  Proportion of participants whose medical billing account is administratively marked as past due within 12 months following baseline
Out of pocket (OOP) expenditures | between baseline and 12 months
  Average OOP expenditures per patient between baseline and 12 months following baseline
Patient Assessment of cancer Communication Experiences (PACE) | between baseline and 12 months
  16-item instrument intended to assess patient perspective on communication over the course of cancer care. The survey items are conceptually grounded in the 6 functions of patient-centered communication: fostering healing relationships, effectively exchanging information, responding to emotions, making quality decisions, managing uncertainty, and enabling patient self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Nora B Henrikson, PhD, MPH, Principal Investigator — Kaiser Permanente; Matthew Banegas, PhD, MPH, MS, Principal Investigator — University of California, San Diego; Amanda Petrik, PhDC, MS, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henrikson NB, Anderson ML, Dickerson J, Petrik AF, Figueroa Gray M, Ewing JJ, Garcia R, Keast E, King DA, Locher B, Scrol A, Ramaprasan A, Rivelli JS, Schneider JL, Banegas MP. Financial Navigation for People Newly Diagnosed With Cancer: Primary Outcomes From the Cancer Financial Experience Randomized Trial. JCO Oncol Pract. 2025 Dec;21(12):1817-1829. doi: 10.1200/OP-25-00874. Epub 2025 Oct 10. PMID 41070850
- [Derived] Henrikson NB, Anderson ML, Dickerson J, Ewing JJ, Garcia R, Keast E, King DA, Lewis C, Locher B, McMullen C, Norris CM, Petrik AF, Ramaprasan A, Rivelli JS, Schneider JL, Shulman L, Tuzzio L, Banegas MP. The Cancer Financial Experience (CAFE) study: randomized controlled trial of a financial navigation intervention to address cancer-related financial hardship. Trials. 2022 May 13;23(1):402. doi: 10.1186/s13063-022-06344-3. PMID 35562781